CLINICAL TRIAL: NCT04964557
Title: A Randomised, Parallel, Double-Blind, Placebo-Controlled Phase 2b Study to Assess the Safety, Tolerability and Efficacy of AZD8233 Treatment in Participants With Hyperlipidaemia
Brief Title: A Study to Assess the Safety, Efficacy and Tolerability of AZD8233 Treatment in Participants With Hyperlipidaemia
Acronym: SOLANO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7990C00004; 2020-005845-18 (EudraCT Number)
Record Dates: First submitted 2021-06-15; First posted 2021-07-16 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-11

CONDITIONS: Hyperlipidaemia
Keywords: AZD8233; Efficacy; PK; PD; Safety; Tolerability
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD8233 (Experimental): AZD8233 for subcutaneous use
  Interventions: Drug: AZD8233
- Placebo (Placebo Comparator): Placebo solution for subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8233 — PCSK9-targeted ASO for the reduction of circulating levels of LDL-C.
  Arms: AZD8233
Drug: Placebo — Placebo solution
  Arms: Placebo

SUMMARY:
AZD8233 is a PCSK9-targeted ASO for the reduction of circulating levels of LDL-C. This study aims to evaluate safety, efficacy and tolerability of AZD8233.

DETAILED DESCRIPTION:
This is a randomized parallel, double-blind, placebo-controlled Phase 2b study in approximately 376 participants with hyperlipidaemia. The primary objective of the study is to assess the safety and tolerability of AZD8233 as compared with placebo, and the effect of AZD8233 versus placebo on relative change in LDL-C. The study will be conducted at up to 100 sites in up to 8 countries.

The screening period starts up to 28 days before the randomization visit and ends on Day -1. Eligible participants will attend 1 enrollment visit and 15 visits during the treatment period and 2 additional visits during the safety follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 75 years of age, inclusive, at the time of signing the informed consent
* Participants who have a fasting LDL-C ≥ 70 mg/dL (1.8 mmol/L) but < 190 mg/dL (4.9 mmol/L) at screening
* Participants who have fasting triglycerides < 400 mg/dL (< 4.52 mmol/L) at screening
* Participants are receiving a stable dose (≥ 3 months) of maximally tolerated statin and/or ezetimibe therapy
* Male or female of non-childbearing potential
* Signed and dated written informed consent prior to any mandatory study specific procedures, sampling, and analyses

Exclusion Criteria:

* eGFR < 40 mL/min/1.73m2 using the CKD-EPI
* History or presence of gastrointestinal, hepatic or renal disease or any other conditions known to interfere with absorption, distribution, metabolism or excretion of drugs
* Any uncontrolled or serious disease, or any medical (eg,. known major active infection or major haematological, renal, metabolic, gastrointestinal or endocrine dysfunction) or surgical condition that, in the opinion of the investigator, may either interfere with participation in the clinical study and/or put the participant at significant risk (according to the investigator's judgment) if he/she participates in the clinical study
* Poorly controlled T2DM, defined as HbA1c > 10%
* Acute ischaemic cardiovascular events including stroke within 30 days, or heart failure with New York Heart Association (NYHA) Class III to IV
* Blood dyscrasias with increased risk of bleeding including idiopathic thrombocytopenic purpura and thrombotic thrombocytopenic purpura or symptoms of increased risk of bleeding (frequent bleeding gums or nose bleeds)
* High-risk of bleeding diathesis or anti-platelet therapy other than low dose aspirin (≤100mg/day).
* Malignancy within the last 10 years
* Recipient of any major organ transplant
* LDL or plasma apheresis within 12 months prior to randomisation
* Uncontrolled hypertension defined as average supine SBP > 160 mmHg or DBP > 90 mmHg
* Heart rate after 10 minutes supine rest < 50 or > 100 bpm
* Any laboratory values with the following deviations at the Screening Visit; test may be repeated at the discretion of the investigator if abnormal:

  * Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV)
  * ALT > 1.5 × ULN
  * AST > 1.5 × ULN
  * TBL > ULN
  * ALP > 1.5 × ULN
  * WBC < lower limit of normal (LLN).
  * Haemoglobin < 12 g/dL in males or < 11 g/dL in females
  * Platelet count ≤ LLN
  * aPTT > ULN or Prothrombin Time > ULN
  * UACR > 11 mg/mmol (100 mg/g)
  * UPCR > 300 mg/g
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG
* QTcF > 470 ms; high degree atrioventricular (AV)-block grade II-III and sinus node dysfunction with significant sinus pause untreated with pacemaker; and cardiac tachyarrhythmias
* History of drug and/or alcohol abuse or a positive screen for drugs of abuse
* Use of warfarin, direct or indirect thrombin inhibitors or factor Xa inhibitors
* Mipomersen, or lomitapide within 12 months prior to randomisation
* Any fibrate therapy other than fenofibrate; if the participant is on fenofibrate therapy, the dose should be stable for at least 6 weeks prior to randomisation
* Previous administration of AZD8233/AZD6615) or inclisiran (LEQVIO ® Novartis)
* Use of evolocumab (REPATHA® Amgen) and alirocumab (PRALUENT® Regeneron) within 3 months of screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (64):
- United States (15):
  - Research Site, Huntsville, Alabama
  - Research Site, Canoga Park, California
  - Research Site, Lincoln, California
  - Research Site, Inverness, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Meridian, Idaho
  - Research Site, Indianapolis, Indiana
  - Research Site, New Windsor, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Stow, Ohio
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Suffolk, Virginia
- Czechia (10):
  - Research Site, Benešov
  - Research Site, Brandýs nad Labem
  - Research Site, Brno
  - Research Site, Jaroměř
  - Research Site, Liberec
  - Research Site, Louny
  - Research Site, Ostrava-Dubina
  - Research Site, Příbram
  - Research Site, Teplice
  - Research Site, Uherské Hradiště
- Denmark (8):
  - Research Site, Aarhus N
  - Research Site, Herlev
  - Research Site, Herning
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Roskilde
  - Research Site, Svendborg
  - Research Site, Viborg
- Hungary (4):
  - Research Site, Balatonfüred
  - Research Site, Békéscsaba
  - Research Site, Debrecen
  - Research Site, Orosháza
- Netherlands (6):
  - Research Site, Amsterdam
  - Research Site, Doetinchem
  - Research Site, Ede
  - Research Site, Gouda
  - Research Site, Harderwijk
  - Research Site, Rotterdam
- Poland (8):
  - Research Site, Bydgoszcz
  - Research Site, Chrzanów
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Puławy
  - Research Site, Ruda Śląska
  - Research Site, Tychy
  - Research Site, Wierzchosławice
- Slovakia (7):
  - Research Site, Bratislava
  - Research Site, Brezno
  - Research Site, Lučenec
  - Research Site, Prešov
  - Research Site, Rožňava
  - Research Site, Svidník
  - Research Site, Trebišov
- Spain (6):
  - Research Site, A Coruña
  - Research Site, Ferrol
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSRsynopsis_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7990C00004&attachmentIdentifier=a87bb6e5-4f84-4af3-a19b-5b24e99a5ec2&fileName=d7990c00004-study-synopsis_(1)_Redacted.pdf&versionIdentifier=
- See also: CSP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7990C00004&attachmentIdentifier=6ba09ee4-0e01-41bd-936b-b22d2fec79ce&fileName=D7990C00004__Protocol_Redacted.pdf&versionIdentifier=
- See also: SAP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7990C00004&attachmentIdentifier=51966def-7e02-40e9-ad3b-c72fa72efdbd&fileName=d7990c00004-sap-ed-4_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a total of 66 study centres in 8 countries: Czech Republic (10 centres), Denmark (8 centres), Hungary (4 centres), Netherlands (6 centres), Poland (8 centres), Slovakia (7 centres), Spain (7 centres), and United States (16 centres). First subject enrolled: 07 July 2021 and Last subject last visit: 15 July 2022.
Groups:
- Placebo: Matching placebo solution for subcutaneous injection.
Period: Overall Study
Arm/Group | AZD8233 | Placebo
Started | 206 | 205
Completed | 196 | 201
Not Completed | 10 | 4
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Death | 3 | 0
Not completed — Reported by investigator as completed but did not fulfil the Completed study definition. | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is based on the Full analysis set (FAS) which includes all subjects who were randomly assigned to study intervention. Subjects were analysed according to their randomised study medication assignment, irrespective of the treatment actually received. Number Started in the Participant Flow is the number of subjects who were randomised.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD8233 | Placebo | Total
Number analyzed (Participants) | 206 | 205 | 411
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (8.1) | 62.2 (7.7) | 62.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 94 | 195
  Male | 105 | 111 | 216
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 2 | 4
  Black or African American | 9 | 3 | 12
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White | 194 | 199 | 393
Region of Enrollment [Number; unit: Participants] — Population: The table contains all subjects randomized (Full analysis set)
  Participants
    USA | 48 | 39 | 87
    Czech Republic | 45 | 44 | 89
    Denmark | 31 | 21 | 52
    Hungary | 15 | 14 | 29
    Netherlands | 12 | 7 | 19
    Poland | 4 | 10 | 14
    Slovakia | 35 | 43 | 78
    Spain | 16 | 27 | 43
LDL-C [Mean (Standard Deviation); unit: mg/dL] — Baseline LDL-C
  mg/dL | 103 (31.8) | 107.4 (31.9) | 105.2 (31.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline on Serum LDL-C
Description: Percentage change in Low-density Lipoprotein Cholesterol (LDL-C) from baseline to Day 197.
Time Frame: From baseline to Day 197
Population: Full analysis set includes all subjects who were randomly assigned to study intervention. Subjects were analysed according to their randomised study medication assignment, irrespective of the treatment actually received.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | AZD8233 | Placebo
Number analyzed (Participants) | 206 | 205
percent change | -56.7 [-60.8 to -52.7] | 5.6 [1.5 to 9.6]
Statistical Analysis 1: Comparison: AZD8233 vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -62.3, 95% CI 2-sided [-68 to -56.6]

2. Secondary Outcome: Percentage Change From Baseline on Serum PCSK9
Description: Percentage change in Proprotein convertase subtilisin/kexin type-9 (PCSK9) from baseline to Day 197.
Time Frame: From baseline to Day 197
Population: Full analysis set includes all subjects who were randomly assigned to study intervention. Subjects will be analysed according to their randomised study medication assignment, irrespective of the treatment actually received.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | AZD8233 | Placebo
Number analyzed (Participants) | 206 | 205
percent change | -77.5 [-81.1 to -74] | -0.8 [-4.3 to 2.6]
Statistical Analysis 1: Comparison: AZD8233 vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -76.7, 95% CI 2-sided [-81.7 to -71.7]

3. Secondary Outcome: Plasma Concentration of AZD8233
Description: AZD8233 full length ASO concentrations in plasma were summarised by descriptive statistics by sampling time point and listed on individual level based on the PK analysis set.
Time Frame: Pre-dose of Day 29, Day 85, Day 141, Day 183, Day 197
Population: The PK analysis set consists of all subjects who receive at least 1 dose of AZD8233, for whom at least 1 post-dose PK concentration assessment is available. Subjects were allocated to the actual treatment received. The number analyzed represents the number of participants with available PK data at that time point, including lower limit of quantification (LLoQ) observations, but not included in the calculation of summary statistics of Geometric Mean and Geometric Coefficient of Variation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AZD8233
Number analyzed (Participants) | 200
ng/mL
  Day 29: number analyzed (Participants) | 195
  Day 29 | 0.2648 (82.8352)
  Day 85: number analyzed (Participants) | 189
  Day 85 | 0.3927 (84.9378)
  Day 141: number analyzed (Participants) | 186
  Day 141 | 0.5749 (161.9301)
  Day 183: number analyzed (Participants) | 171
  Day 183 | 1.0441 (178.5196)
  Day 197: number analyzed (Participants) | 185
  Day 197 | 0.6975 (208.2431)

4. Secondary Outcome: Anti-drug Antibodies (ADAs) During the Treatment Period and Follow-up Period
Description: Number of ADA positive subjects at each time point during the treatment period and follow-up period.
Time Frame: Pre-dose of Day 1, Day 29, Day 57, Day 85, Day 113, Day 141, Day 169, Day 197, Day 281
Population: The safety analysis set consists of all subjects who have received at least one dose of investigational product. Erroneously treated subjects (e.g., those randomised to treatment A but actually given treatment B) are accounted for in the treatment group of the treatment they actually received. The number analyzed represents the number of participants with available ADA data at that time point.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD8233 | Placebo
Number analyzed (Participants) | 207 | 203
Participants
  Day 1 | 6 | 4
  Day 29: number analyzed (Participants) | 198 | 197
  Day 29 | 15 | 3
  Day 57: number analyzed (Participants) | 196 | 195
  Day 57 | 16 | 3
  Day 85: number analyzed (Participants) | 195 | 198
  Day 85 | 18 | 3
  Day 113: number analyzed (Participants) | 193 | 191
  Day 113 | 21 | 3
  Day 141: number analyzed (Participants) | 188 | 195
  Day 141 | 25 | 2
  Day 169: number analyzed (Participants) | 190 | 193
  Day 169 | 31 | 2
  Day 197: number analyzed (Participants) | 189 | 194
  Day 197 | 37 | 3
  Day 281: number analyzed (Participants) | 185 | 188
  Day 281 | 40 | 3

5. Primary Outcome: Number of Subjects With Adverse Events (AEs)
Description: Please refer to the adverse event module for specifics.
Time Frame: On-study includes adverse events with an onset date on or after the date of first dose of IP through study competition, planned visit date Day 281.
Population: The safety analysis set consists of all subjects who have received at least one dose of investigational product. Erroneously treated subjects (e.g., those randomised to treatment A but actually given treatment B) are accounted for in the treatment group of the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD8233 | Placebo
Number analyzed (Participants) | 207 | 203
Participants | 141 | 127

6. Primary Outcome: Vital Signs - Temperature
Description: Mean and standard deviation of Temperature at each scheduled visit by treatment.
Time Frame: Baseline, Days 15, 29, 57, 85, 113, 141, 169, 197, 225, and 281.
Population: Safety analysis set, the number analyzed represents the number of participants with available temperature data at that time point.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | AZD8233 | Placebo
Number analyzed (Participants) | 207 | 203
Celsius
  Baseline | 36.434 (0.437) | 36.369 (0.389)
  Day 15: number analyzed (Participants) | 201 | 202
  Day 15 | 36.344 (0.404) | 36.387 (0.378)
  Day 29: number analyzed (Participants) | 201 | 198
  Day 29 | 36.360 (0.422) | 36.361 (0.386)
  Day 57: number analyzed (Participants) | 199 | 198
  Day 57 | 36.340 (0.420) | 36.396 (0.368)
  Day 85: number analyzed (Participants) | 195 | 198
  Day 85 | 36.360 (0.416) | 36.362 (0.363)
  Day 113: number analyzed (Participants) | 195 | 194
  Day 113 | 36.359 (0.391) | 36.399 (0.348)
  Day 141: number analyzed (Participants) | 189 | 195
  Day 141 | 36.335 (0.398) | 36.373 (0.341)
  Day 169: number analyzed (Participants) | 194 | 194
  Day 169 | 36.304 (0.454) | 36.353 (0.411)
  Day 197: number analyzed (Participants) | 191 | 195
  Day 197 | 36.299 (0.477) | 36.352 (0.316)
  Day 225: number analyzed (Participants) | 190 | 192
  Day 225 | 36.327 (0.472) | 36.365 (0.37)
  Day 281: number analyzed (Participants) | 186 | 188
  Day 281 | 36.353 (0.396) | 36.391 (0.363)

7. Primary Outcome: Vital Sign - Weight
Description: Mean and standard deviation of Weight at each scheduled visit by treatment.
Time Frame: Baseline and Day 281.
Population: Safety analysis set, the number analyzed represents the number of participants with available weight data at that time point.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | AZD8233 | Placebo
Number analyzed (Participants) | 207 | 203
kg
  Baseline | 86.642 (17.054) | 88.750 (17.566)
  Day 281: number analyzed (Participants) | 183 | 188
  Day 281 | 85.493 (16.561) | 88.759 (18.110)

8. Primary Outcome: Number of Participants With an ECG Determined to be Abnormal and Clinically Significant
Description: Number of participants With an ECG Determined to be Abnormal and Clinically Significant at each scheduled visit by treatment
Time Frame: Baseline, Days 85, 169, 225, and 281.
Population: Safety analysis set, the number analyzed represents the number of participants with available ECG data at that time point.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD8233 | Placebo
Number analyzed (Participants) | 207 | 203
Participants
  Baseline | 0 | 0
  Day 85: number analyzed (Participants) | 190 | 191
  Day 85 | 1 | 1
  Day 169: number analyzed (Participants) | 193 | 193
  Day 169 | 0 | 0
  Day 225: number analyzed (Participants) | 190 | 191
  Day 225 | 0 | 0
  Day 281: number analyzed (Participants) | 185 | 188
  Day 281 | 0 | 0

9. Primary Outcome: Vital Sign - Systolic Blood Pressure
Description: Mean and standard deviation of Systolic Blood Pressure at each scheduled visit by treatment.
Time Frame: Baseline, Days 15, 29, 57, 85, 113, 141, 169, 197, 225, and 281.
Population: Safety analysis set, the number analyzed represents the number of participants with available systolic blood pressure data at that time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD8233 | Placebo
Number analyzed (Participants) | 207 | 203
mmHg
  Baseline | 130.918 (13.284) | 131.325 (11.281)
  Day 15: number analyzed (Participants) | 201 | 202
  Day 15 | 130.438 (13.541) | 131.198 (12.711)
  Day 29: number analyzed (Participants) | 201 | 198
  Day 29 | 130.741 (13.363) | 133.152 (11.881)
  Day 57: number analyzed (Participants) | 199 | 198
  Day 57 | 130.754 (12.536) | 131.465 (14.073)
  Day 85: number analyzed (Participants) | 195 | 198
  Day 85 | 131.913 (12.083) | 132.111 (12.238)
  Day 113: number analyzed (Participants) | 195 | 194
  Day 113 | 131.974 (12.622) | 132.493 (12.022)
  Day 141: number analyzed (Participants) | 189 | 195
  Day 141 | 131.386 (14.246) | 132.041 (14.081)
  Day 169: number analyzed (Participants) | 194 | 194
  Day 169 | 130.959 (11.874) | 132.706 (12.481)
  Day 197: number analyzed (Participants) | 191 | 195
  Day 197 | 129.351 (14.236) | 133.149 (11.838)
  Day 225: number analyzed (Participants) | 190 | 192
  Day 225 | 131.188 (14.578) | 133.165 (12.746)
  Day 281: number analyzed (Participants) | 186 | 188
  Day 281 | 130.048 (13.288) | 131.043 (13.069)

10. Primary Outcome: Vital Sign - Diastolic Blood Pressure
Description: Mean and standard deviation of Diastolic Blood Pressure at each scheduled visit by treatment.
Time Frame: Baseline, Days 15, 29, 57, 85, 113, 141, 169, 197, 225, and 281.
Population: Safety analysis set, the number analyzed represents the number of participants with available diastolic blood pressure data at that time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AZD8233 | Placebo
Number analyzed (Participants) | 207 | 203
mmHg
  Baseline | 78.937 (7.608) | 78.562 (6.134)
  Day 15: number analyzed (Participants) | 201 | 202
  Day 15 | 78.318 (8.060) | 78.559 (6.946)
  Day 29: number analyzed (Participants) | 201 | 198
  Day 29 | 78.408 (8.157) | 79.611 (6.779)
  Day 57: number analyzed (Participants) | 199 | 198
  Day 57 | 78.714 (7.799) | 79.369 (7.120)
  Day 85: number analyzed (Participants) | 195 | 198
  Day 85 | 78.867 (8.053) | 79.081 (7.575)
  Day 113: number analyzed (Participants) | 195 | 194
  Day 113 | 79.164 (8.393) | 79.584 (7.152)
  Day 141: number analyzed (Participants) | 189 | 195
  Day 141 | 78.698 (8.505) | 78.836 (7.758)
  Day 169: number analyzed (Participants) | 194 | 194
  Day 169 | 78.139 (8.489) | 78.402 (7.359)
  Day 197: number analyzed (Participants) | 191 | 195
  Day 197 | 78.382 (7.736) | 78.615 (7.432)
  Day 225: number analyzed (Participants) | 190 | 192
  Day 225 | 78.582 (8.313) | 78.988 (7.254)
  Day 281: number analyzed (Participants) | 186 | 188
  Day 281 | 78.812 (8.484) | 78.601 (7.249)

11. Primary Outcome: Vital Sign - Pulse Rate
Description: Mean and standard deviation of Pulse rate at each scheduled visit by treatment.
Time Frame: Baseline, Days 15, 29, 57, 85, 113, 141, 169, 197, 225, and 281.
Population: Safety analysis set, the number analyzed represents the number of participants with available pulse rate data at that time point.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | AZD8233 | Placebo
Number analyzed (Participants) | 207 | 203
beats/min
  Baseline | 68.93 (11.52) | 67.88 (10.47)
  Day 15: number analyzed (Participants) | 201 | 202
  Day 15 | 70.63 (10.07) | 69.48 (10.42)
  Day 29: number analyzed (Participants) | 201 | 198
  Day 29 | 68.52 (9.91) | 68.90 (10.05)
  Day 57: number analyzed (Participants) | 199 | 198
  Day 57 | 69.58 (10.59) | 69.90 (11.56)
  Day 85: number analyzed (Participants) | 195 | 198
  Day 85 | 68.90 (9.87) | 69.53 (11.10)
  Day 113: number analyzed (Participants) | 195 | 194
  Day 113 | 70.77 (10.58) | 70.03 (10.48)
  Day 141: number analyzed (Participants) | 189 | 194
  Day 141 | 70.85 (11.10) | 70.00 (10.84)
  Day 169: number analyzed (Participants) | 194 | 194
  Day 169 | 69.35 (10.44) | 68.38 (10.31)
  Day 197: number analyzed (Participants) | 191 | 195
  Day 197 | 70.69 (12.26) | 69.43 (8.94)
  Day 225: number analyzed (Participants) | 190 | 192
  Day 225 | 69.56 (10.17) | 68.79 (10.48)
  Day 281: number analyzed (Participants) | 186 | 188
  Day 281 | 68.39 (9.99) | 69.31 (10.90)

12. Primary Outcome: Treatment Emergent Platelet Count Abnormalities
Description: Treatment emergent platelet count abnormalities by pre-specified criteria by treatment.
Time Frame: Treatment emergent includes results after the first dose of IP through study competition, planned visit date Day 281.
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | AZD8233 | Placebo
Number analyzed (Participants) | 207 | 203
Participants
  Platelet count < LLN: number analyzed (Participants) | 206 | 203
  Platelet count < LLN | 9 | 11
  Platelet count > ULN: number analyzed (Participants) | 206 | 203
  Platelet count > ULN | 26 | 20
  Platelet count < 50 x 10^9/L: number analyzed (Participants) | 206 | 203
  Platelet count < 50 x 10^9/L | 0 | 0
  Platelet count < 75 x 10^9/L: number analyzed (Participants) | 206 | 203
  Platelet count < 75 x 10^9/L | 1 | 1
  Platelet count < 100 x 10^9/L: number analyzed (Participants) | 206 | 203
  Platelet count < 100 x 10^9/L | 2 | 2
  Platelet count < 150 x 10^9/L: number analyzed (Participants) | 206 | 203
  Platelet count < 150 x 10^9/L | 19 | 21
  >30% decrease from baseline: number analyzed (Participants) | 206 | 203
  >30% decrease from baseline | 14 | 14
  <150 x 10^9/L or >30% decrease from baseline: number analyzed (Participants) | 206 | 203
  <150 x 10^9/L or >30% decrease from baseline | 28 | 26
  <150 x 10^9/L and >30% decrease from baseline: number analyzed (Participants) | 206 | 203
  <150 x 10^9/L and >30% decrease from baseline | 5 | 9

ADVERSE EVENTS:
Time Frame: On-study includes adverse events with an onset date on or after the date of first dose of IP through study competition, planned visit date Day 281.
Description: The safety analysis set consists of all subjects who have received at least one dose of investigational product. Erroneously treated subjects (e.g., those randomised to treatment A but actually given treatment B) are accounted for in the treatment group of the treatment they actually received.
Arm/Group | AZD8233 | Placebo
All-Cause Mortality (participants affected / at risk) | 3/207 | 0/203
Serious Adverse Events (participants affected / at risk) | 18/207 | 12/203
Other Adverse Events (participants affected / at risk) | 69/207 | 62/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8233 (N=207) | Placebo (N=203)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2)
Sudden death (General disorders) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Coagulation time prolonged (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma urethra (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Bipolar i disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8233 (N=207) | Placebo (N=203)
Injection site reaction (General disorders) | 22 (56) | 5 (7)
Covid-19 (Infections and infestations) | 33 (33) | 36 (37)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 18 (19) | 14 (14)
Hypertension (Vascular disorders) | 11 (11) | 13 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT04964557/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT04964557/SAP_001.pdf